CLINICAL TRIAL: NCT03829813
Title: Does Music Therapy Improve Patient Mood, Pain, Satisfaction and Caregiver Satisfaction on Adult Inpatient Acute Neurological Units?
Brief Title: Effects of Music Therapy on Mood, Pain, Patient and Staff Satisfaction on Adult Inpatient Neurological Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: National Music Centre Studio Bell (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB18-1145
Record Dates: First submitted 2018-10-26; First posted 2019-02-04 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2018-10

CONDITIONS: Music Therapy; Pain; Patient Satisfaction; Inpatients; Affect
MeSH Terms: conditions — Pain; Patient Satisfaction | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Mixed methods study with pre and post intervention surveys and Visual analog scales, combined with focus groups/interviews of patients, family members and staff
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients (Experimental): Music therapy sessions. Planned 1:1 within acute neurology/rehabilitation patient rooms, or private rooms by a qualified music therapist once weekly and/or group music therapy sessions maximum 6-8 patients for less than or equal to one hour. Music therapy includes a variety of techniques used to target mood, pain, socialisation, expressive speech, attention/cognitive or sensorimotor functional goals.
  Interventions: Other: Music therapy
- Family (Experimental): Family participation in music therapy treatment sessions. Planned 1:1 within acute neurology/rehabilitation patient rooms, or private rooms by a qualified music therapist once weekly and/or group music therapy sessions maximum 6-8 patients for less than or equal to one hour.
  Interventions: Other: Music therapy
- Administration and Staff (Experimental): Staff/Administration are not participants in music therapy, but rather have observed sessions, or worked as co-treating clinicians with music therapists for patient participants.
  Interventions: Other: Music therapy

INTERVENTIONS:
Other: Music therapy — 20 to 40 minute music therapy treatment session with a qualified music therapist.

SUMMARY:
A study examining the benefits of music therapy on patients, families, and unit staff on acute neurologic or inpatient rehabilitation units.

DETAILED DESCRIPTION:
Objective: Does music therapy improve mood, pain and patient satisfaction on adult inpatient neurological units? Is music therapy an acceptable and feasible intervention in an adult inpatient neurological unit based on patient, family, and care provider satisfaction measures?

Population: Foothills Medical Centre (FMC) acute neurological and neurorehabilitation units (i.e., 111, 112, 101, 58 Neurorehab), ages >18

Background: Music therapy is the therapeutic application of music to rehabilitate cognitive, motor, and sensory dysfunction due to disease. Its treatment techniques are based upon scientific knowledge of music perception, production and its effects on nonmusical brain and behavior functions like gait, balance, speech, mood and motivation. Music is also known to have a wide range of physiological effects on the human body including changes in heart rate, respiration, blood pressure, skin temperature, and muscle tension. Music provokes emotions mediated via neuro-hormones such as serotonin and dopamine, and is experienced as joyous or rewarding through activity changes in the amygdala, ventral striatum and other parts of the limbic system.

Music therapy has been applied across a broad range of clinical conditions from inpatients to outpatients, cardiac, diabetes and cancer care to surgical and ICU settings, and in pediatric through adult and geriatric populations. The majority of clinical studies focus on neurological patients with sensorimotor, speech and gait impairments, however, music has been shown to improve mental state and functioning in a wide variety of psychiatric disorders including depression, anxiety, and dementia, as well as reducing anxiety in patients with asthma, osteoarthritis, those undergoing dental procedures or perioperative anesthesia. There is some research to support its mood benefits in stroke and brain injury patients.

Music therapy has been found to be an effective complementary treatment for cancer-related pain, lithotripsy, labor, and fibromyalgia. Recent reviews have demonstrated reductions in postoperative pain and anxiety, decreased consumption of sedatives and analgesics and increased patient satisfaction. The reductions in anxiety were equal or greater than midazolam/benzodiazepines. This may be particularly beneficial in neurological patients who may be more susceptible to adverse effects from psychoactive, sedating and analgesic medications. Music can provide a filter for unpleasant, unfamiliar sounds common to the hospital environment and improve sleep quality. These positive effects may greatly assist the common issues of fatigue in cognitively impaired, confused or agitated neurological inpatients. Furthermore, Chlan has recently demonstrated cost-effectiveness of music therapy interventions in reducing anxiety in the ICU.

Music therapy may also have beneficial effects for staff and families. Some studies have demonstrated cost-effectiveness with less staff time required for procedures, administering sedatives and pain medications, and fewer days on mechanical ventilation in the ICU. Perez-Cruz studied patients, relatives, and healthcare workers' preference for background music in patient areas with an average 71% in all three groups. Lower perceived stress level, cortisol, heart rate and mean arterial pressures were also observed in voluntary first-line nurses and students while listening to music.

This study will expand the research base in the inpatient neurological population and explore staff perceptions and satisfaction with music therapy. The aim of this mixed methods study is to explore immediate pre and post music therapy intervention effects on mood, pain, and satisfaction in the inpatient neurological population and to explore perceived caregiver and staff satisfaction with music therapy on inpatient neurological units.

Intervention: 20-40 min treatment sessions 1:1 within acute neurological patient rooms, or private room by qualified music therapist once weekly and/or group music therapy sessions maximum 6-8 patients < or = 1 hour. This includes a variety of music therapy techniques used to target mood, pain, socialization, expressive speech, attention/cognitive or sensorimotor functional goals.

Methods: Mixed methods study design.

1. Qualitative measures:

   1. Semi-structured patient +/- family satisfaction questionnaire and interview post music therapy session
   2. Semi-structured inpatient unit staff questionnaire and interview (exploring themes of: self-perceived stress, workload, barriers, relationships, mood, pain)
   3. Focus groups of patients, families, staff addressing above areas
2. Quantitative measures:

   1. Visual analog scale, mood pre- and post- music therapy session
   2. Visual analog scale, pain pre- and post- music therapy session

Recruitment: Patients (and their families when available) referred to Music therapy on Acute Neuro, Neurorehab units would be invited to participate in research study with informed consent obtained prior to interviews, focus groups and data collection. Unit Staff would also be invited to participate in interviews and focus groups with informed consent prior to data collection.

ELIGIBILITY:
Inclusion Criteria:

* Acute neurological inpatients and their families at Foothills Medical Centre that are receiving music therapy
* Unit staff involved in care of patients receiving music therapy as inpatients
* Age > 18

Exclusion Criteria:

* Non-English speaking participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Qualitative data from focus groups | Up to 1 month following music therapy intervention
  Questions within the interview are designed to more deeply explore the areas of music therapy and how this program may influence stress, mood, pain, and the relationships between participants, caregivers, and hospital staff. Interviews will also touch upon barriers to music therapy involvement as experienced.

SECONDARY OUTCOMES:
Pain Visual Analogue Scale | T0 (prior to music therapy treatment, T(1) immediately following music therapy treatment
  Measurement instrument that measures participants subjective perception of pain believed to range across a continuum of values.
  Scale: 0 (minimum, no pain) - 10 (maximum, very severe pain).
Mood Visual Analogue Scale | T0 (prior to music therapy treatment, T(1) immediately following music therapy treatment
  0 (minimum, not at all happy) - 10 (maximum, very happy).
Patient Satisfaction | T0 (prior to music therapy treatment, T(1) immediately following music therapy treatment
  Likert Scale:
  1. - Very dissatisfied
  2. - Somewhat dissatisfied
  3. - Neutral
  4. - Somewhat satisfied
  5. - Very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Plamondon, Principal Investigator — University of Calgary
Locations (1):
- Foothill Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No